CLINICAL TRIAL: NCT00727389
Title: The Influence of the Support Group on the Functional Incapacity in the Prevention of Functional Decline of Aged Women.
Brief Title: Prevention of Functional Decline of Aged Women
Acronym: Incapacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Cearense de Odontologia (Other)
Collaborators: Fortaleza University (Other)
Responsible Party: Maria Vieira de Lima Saintrain, Universidade de Fortaleza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: lnunes
Record Dates: First submitted 2008-07-28; First posted 2008-08-04 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Health Care Quality, Access, and Evaluation
Keywords: Prevention; Quality of Health Care; Health Care Evaluation Mechanisms
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- groups of women (Other): To evaluate the capacity of muscular function and articular amplitude in the aged women
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Physiotherapy — Exercise two days a week for six month
  Other Names: muscle function; articular amplitude

SUMMARY:
The objective of this study is to evaluate the capacity of muscular function and articular amplitude in the aged women who participated in the Support Group and its influence on the prevention of function decline of these women.

DETAILED DESCRIPTION:
To evaluate the capacity of muscular function and articular amplitude in the aged women who participated the Support Group and its influence on the prevention of function decline of these women is use the method: It is an interventional and quantitative research. A questionnaire of identification and instruments will use: a) flexion and extension tests of muscular function and articular amplitude of shoulders, elbows, wrists, hip, knees and ankles, in the beginning and in the end of the program b) educational action c) physical exercise d) the check up of the results after the exercises e) two questions to register the influence of the support group in the functional life of the researched ones.

ELIGIBILITY:
Inclusion Criteria:

* woman with 60 years old or more

Exclusion Criteria:

* woman with less 60 years old

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
A instrument was used for flexion and extension tests of muscular function and articular amplitude of shoulders, elbows, wrists, hip, knees and ankles, in the beginning and in the end of the program; physical exercise; the check up of the results | six month

CONTACTS AND LOCATIONS:
Overall Officials: Maria VL Saintrain, doutor, Study Director — Universidade de Fortaleza
Locations (1):
- Grupo de apoio a prevenção da incapacidade funcional, Fortaleza, Ceará, Brazil